CLINICAL TRIAL: NCT00005352
Title: Chronic Stress as a Risk Factor in the Etiology of Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4231; R01HL047325 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To conduct a prospective, longitudinal, analysis of the psychophysiological effects of chronic exposure to environmental stress. The study took advantage of a unique, naturally occurring experiment caused by the relocation of a major international airport.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Studies were conducted on blood pressure and the neuroendocrine effects of noise resulting from the relocation of the Munich International Airport. At the former airport site the investigators monitored people exposed to high levels of noise and then tracked these same individuals as their ambient environment became normal following the shutdown of the airport. At the new airport site, the opposite situation occurred: Individuals living in normal, quiet ambient conditions became exposed to loud aircraft noise. At both sites, control groups were formed who were not exposed to aircraft noise. The study piggybacked onto a German sponsored grant. NIH funds covered the costs of cardiovascular and psycho-physiological data analysis. Measures included biochemical assays of chronic neuroendocrine markers of stress, resting blood pressure, and reactivity of blood pressure during cognitive tasks. Perceptions of community noise levels were also assessed as possible mediators of the stressful effects of chronic exposure to ambient, environmental noise.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1996-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Evans — Cornell University

REFERENCES:
- [Background] Tafalla RJ, Evans GW. Noise, physiology, and human performance: the potential role of effort. J Occup Health Psychol. 1997 Apr;2(2):148-55. doi: 10.1037//1076-8998.2.2.148. PMID 9552287
- [Background] Bullinger M, Hygge S, Evans GW, Meis M, von Mackensen S. The psychological cost of aircraft noise for children. Zentralbl Hyg Umweltmed. 1999 Aug;202(2-4):127-38. PMID 10507123
- [Background] Hygge S, Evans GW, Bullinger M. A prospective study of some effects of aircraft noise on cognitive performance in schoolchildren. Psychol Sci. 2002 Sep;13(5):469-74. doi: 10.1111/1467-9280.00483. PMID 12219816